CLINICAL TRIAL: NCT01251419
Title: The Impact of Social Proximity on Conversion to Generic Prescription Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 0002; P30AG034532 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Conversion From Brand Name to Generic Medication
Keywords: Generic Medication; Brand Name Medication; Conversion Rates; Social Proximity; Behavioral Economics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Testimonial and Union Arm (Experimental): The testimonial and union arm will receive the same letter as the testimonial treatment arm but with the addition of the union affiliation of the employee giving the testimonial.
  Interventions: Other: Social Proximity and Conversion to Generic Medications
- Control (Experimental): The control arm will receive a letter signed by our partner company's Chief Medical Officer, explaining the health and monetary benefits of switching from brand name prescription medication to generic prescription medication.
  Interventions: Other: Social Proximity and Conversion to Generic Medications
- Testimonial Treatment Arm (Experimental): The testimonial treatment arm will receive the exact same letter as the control arm, but the letter will feature an employee's testimonial along with the first name, last initial, city and state of the employee giving the testimonial.
  Interventions: Other: Social Proximity and Conversion to Generic Medications

INTERVENTIONS:
Other: Social Proximity and Conversion to Generic Medications — At companies where employees are predominantly union members, we will compare the efficacy of a peer information intervention using a testimonial from a union identified employee to an intervention using a testimonial with no union identification, as well as to a no-testimonial intervention.

SUMMARY:
The goal of this project is to understand the effects of receiving peer information on individuals' conversion rates from brand name prescription medication to generic prescription medication.

DETAILED DESCRIPTION:
At companies where employees are predominantly union members, we will compare the efficacy of a peer information intervention using a testimonial from a union identified employee to an intervention using a testimonial with no union identification, as well as to a no-testimonial intervention.

The control arm will receive a letter signed by our partner company's Chief Medical Officer, explaining the health and monetary benefits of switching from brand name prescription medication to generic prescription medication. The testimonial treatment arm will receive the exact same letter, but the letter will feature an employee's testimonial along with the first name, last initial, city and state of the employee giving the testimonial. The testimonial and union arm will receive the same letter as the testimonial treatment arm but with the addition of the union affiliation of the employee giving the testimonial.

ELIGIBILITY:
Inclusion Criteria:

* Employee of a company that uses Express Scripts as its pharmacy benefits manager.
* Employee at a company with predominantly union employees.
* Currently taking a brand name medication with an exact generic equivalent.

Exclusion Criteria:

* Employees on any psychological prescription medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Actual)
Dates: Start 2011-03; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Conversion from Brand Name to Generic Prescription Medication | One month to one year after the intervention.
  We will measure conversion rates of employees from brand name to generic prescription medication by treatment arm.

SECONDARY OUTCOMES:
Union Status and Conversation to Generic Medication | One month to one year after the intervention.
  We will see how union affiliation affects the employee conversion rates from brand name to prescription medication by treatment arm.

CONTACTS AND LOCATIONS:
Overall Officials: David Laibson, Ph.D, Principal Investigator — National Bureau of Economic Research
Locations (1):
- Express Scripts, St Louis, Missouri, United States